CLINICAL TRIAL: NCT06589011
Title: Postoperative Hypoxemia in Obese Patients: Pressure Support Versus Spontaneous Ventilation During Anesthetic Emergence in Laparoscopic Bariatric Surgery: A Randomized Controlled Trial
Brief Title: Postoperative Hypoxemia in Obese Patients
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, lecturer of anesthesia and intensive care medicine, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PT(735); PT(735) (Registry Identifier: TBRI (REC) (FWA#000010609)); (FWA#000010609) (Registry Identifier: Research Ethics Committee (REC))
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Atelectasis, Postoperative Pulmonary; Bariatric Surgery
Keywords: pressure support; postoperative atelectasis; obese patients; bariatric surgery
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: pressure support versus spontaneous assisted ventilation during extubation from bariatric surgeries.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure support (Active Comparator): The initial pressure support ventilation setting was a driving pressure of 7 cm H2O, PEEP of 5 cm H2O, and safety backup ventilation of 12 breaths/min (safety backup ventilation setting, VT, 8 ml/kg of predicted body weight; and PEEP, 5 cm H2O). The flow trigger and end of breath were set at 2 l/min and 30% of peak flow, respectively.
  Interventions: Other: Pressure Support Ventilation
- control group (Placebo Comparator): The emergence process was led by the discretion of the attending anesthesiologist. The basic strategy was to allow the patient to breathe spontaneously and only help respiration if necessary, with intermittent manual assistance.
  Interventions: Other: spontaneously assisted breathing

INTERVENTIONS:
Other: Pressure Support Ventilation — The initial pressure support ventilation setting was a driving pressure of 7 cm H2O, PEEP of 5 cm H2O, and safety backup ventilation of 12 breaths/min
  Arms: Pressure support
Other: spontaneously assisted breathing — The basic strategy was to allow the patient to breathe spontaneously and only help respiration if necessary, with intermittent manual assistance.
  Arms: control group

SUMMARY:
Postoperative atelectasis can cause postoperative hypoxia which might be avoided by applying pressure support during extubation of obese patients undergoing bariatric surgeries.

DETAILED DESCRIPTION:
Postoperative atelectasis is one of the most common pulmonary complications in surgical patients, and a fair majority of studies have suggested that postoperative atelectasis is harmful. It increases the risk of hypoxemia and forms the pathophysiologic basis for other postoperative pulmonary complications. Atelectasis can last for several days after surgery impairing respiratory function, and ultimately delaying patient discharge.

Obese patients are more likely than non-obese patients to develop atelectasis that resolves more slowly. This is because of a marked impairment of the respiratory mechanics (decreased chest wall and lung compliance and decreased functional residual capacity) promoting airway closure with reduction of the oxygenation index (Pao2/ PAo2) to a greater extent than in healthy-weight +subjects . Also the weight of the abdomen makes diaphragmatic excursions more difficult, especially when recumbent or supine, which is intensified in the setting of diaphragmatic paralysis associated with neuromuscular blockade.

Although there have been many studies regarding ventilatory techniques to reduce postoperative pulmonary complications, only a few studies have focused on the period of recovery from anesthesia. The benefits obtained from the protective ventilation techniques may be lost during this emergence process. Whalen et al. found that recruitment maneuver and the application of positive end-expiratory pressure (PEEP) improved intraoperative oxygenation, but the effect dissipated promptly after extubation. Many studies have observed the development of atelectasis during the emergence period. Furthermore, it is estimated that the emergence period contributes to approximately 39% of the total amount of postoperative atelectasis.

Currently, we allow patients to breathe spontaneously and assist their respiration intermittently during the transition from controlled ventilation to spontaneous respiration while assessing whether the patients have enough power to breathe without assistance. However, patients who are spontaneously breathing remain under the influence of residual anesthetic agents and neuromuscular blockers and may not have restored their functional residual capacity, subsequently developing atelectasis. In addition, pain-induced respiratory restriction or respiratory muscle fatigue during spontaneous respiration may increase the risk of atelectasis.

Pressure support ventilation is widely used for weaning from mechanical ventilation in the intensive care unit (ICU) and is recently available in anesthesia machines. Pressure support ventilation applies a fixed amount of pressure the physician selects to the patients throughout each breath to augment their own respiration and is one of the most comfortable ventilation modes for patients. In these aspects, pressure support ventilation during recovery from anesthesia may reduce postoperative atelectasis compared to spontaneous respiration with intermittent manual assistance. To date, few studies have assessed the effect of pressure support ventilation on postoperative atelectasis.

Moreover, laparoscopic surgery are associated with a higher risk of postoperative atelectasis due to the high intra-abdominal pressure which pushes the diaphragm upward and subsequently results in the collapse of the alveoli.

Our hypothesis is that pressure support ventilation will reduces the postoperative hypoxemia and atelectasis compared to spontaneous respiration with intermittent manual assistance during anesthetic emergence in obese patients undergoing laparoscopic surgery.

Aim of the study:

The aim of our study is to assess the possible superiority of pressure support ventilation compared to spontaneous respiration with intermittent manual assistance to reduce postoperative hypoxemia and atelectasis during anesthetic emergence in obese patients undergoing laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-III patients.
2. aged from 18-60 years old.
3. body mass index :(BMI) ≥ 35 Kg/m2 scheduled for laparoscopic bariatric surgery.

Exclusion Criteria:

1. age ≤18 or ≥ 60 years.
2. pregnant females.
3. underlying lung pathology, moderate to severe impairment of RFT, previous lung surgery, pneumothorax and pleural effusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
arterial Pao2 | immediately after arrival to the PACU within 10 minutes after extubation.
  Arterial blood sample was with drawn from the patients on room air after extubation

SECONDARY OUTCOMES:
Postoperative atelectasis | 30 minutes after arrival to the PACU
  diagnosed by chest x-ray
respiratory rescue measures | within 48 hours postoperatively
  need for oxygen supplementation or mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Moshira Sayed Lecturer of anesthesia and intensive care, M.D., Principal Investigator — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research institute, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be available upon request from the principal investigator

REFERENCES:
- [Background] Young CC, Harris EM, Vacchiano C, Bodnar S, Bukowy B, Elliott RRD, Migliarese J, Ragains C, Trethewey B, Woodward A, Gama de Abreu M, Girard M, Futier E, Mulier JP, Pelosi P, Sprung J. Lung-protective ventilation for the surgical patient: international expert panel-based consensus recommendations. Br J Anaesth. 2019 Dec;123(6):898-913. doi: 10.1016/j.bja.2019.08.017. Epub 2019 Oct 3. PMID 31587835
- [Background] van Kaam AH, Lachmann RA, Herting E, De Jaegere A, van Iwaarden F, Noorduyn LA, Kok JH, Haitsma JJ, Lachmann B. Reducing atelectasis attenuates bacterial growth and translocation in experimental pneumonia. Am J Respir Crit Care Med. 2004 May 1;169(9):1046-53. doi: 10.1164/rccm.200312-1779OC. Epub 2004 Feb 20. PMID 14977624
- [Background] Jeong H, Tanatporn P, Ahn HJ, Yang M, Kim JA, Yeo H, Kim W. Pressure Support versus Spontaneous Ventilation during Anesthetic Emergence-Effect on Postoperative Atelectasis: A Randomized Controlled Trial. Anesthesiology. 2021 Dec 1;135(6):1004-1014. doi: 10.1097/ALN.0000000000003997. PMID 34610099